CLINICAL TRIAL: NCT07360834
Title: Predicting Cancer Onset in Lynch Syndrome by Liquid Biopsies
Brief Title: Study Aiming to Test Whether Non-invasive Liquid Biopsies Can Safely Reduce Invasive Surveillance Methods in Lynch Syndrome
Acronym: PREDI-LYNCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UC-GIG-2522; Project 101213916 (Other Grant/Funding Number: EUROPEAN HEALTH AND DIGITAL EXECUTIVE AGENCY (HADEA))
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Lynch Syndrome
Keywords: Lynch Syndrome, hereditary cancer, MMR deficiency, Liquid biopsies, cancer early detection.; Lynch Syndrome, MMR deficiency, Liquid biopsies
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Turcot syndrome | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Biopsies Liquids +/- Colonoscopy
  Interventions: Diagnostic Test: INVITRO DIAGNOSTIC TESTS AND COLONOSCOPY
- Control arm (Other): Colonoscopy each 18 months
  Interventions: Diagnostic Test: INVITRO DIAGNOSTIC TESTS AND COLONOSCOPY

INTERVENTIONS:
Diagnostic Test: INVITRO DIAGNOSTIC TESTS AND COLONOSCOPY — The trial compares two strategies: standard follow-up with colonoscopy every 18 months versus an approach combining annual liquid biopsies with a colonoscopy every 36 months

SUMMARY:
Lynch syndrome is an inherited genetic predisposition that increases the risk of developing several types of cancer, particularly colon and rectal cancers (colorectal cancer), as well as cancer of the uterine lining (endometrial cancer). It affects around 1 in 400 people in Europe.

Today, surveillance mainly relies on examinations such as colonoscopy (an examination of the colon using a camera) or gynaecological evaluations, sometimes accompanied by biopsies (the removal of a small tissue sample for microscopic analysis). Although effective, these procedures are invasive and demanding; they can affect quality of life and discourage some individuals from adhering to their recommended surveillance programme.

The European project PREDI-LYNCH is exploring an additional pathway that is simpler and better tolerated. This project relies on "liquid biopsies", meaning tests performed on easily collected samples such as blood, urine, stool, and vaginal swabs for women with a uterus. The PREDI-LYNCH study aims to determine whether these non-invasive tests could enable personalised surveillance and potentially increase the interval between more burdensome procedures, while maintaining a high level of medical safety.

DETAILED DESCRIPTION:
This European clinical study evaluates whether non-invasive liquid biopsy tests (blood, urine, stool and vaginal samples when applicable) can improve cancer surveillance in adults with genetically confirmed Lynch syndrome (MLH1, MSH2, MSH6 or EPCAM). The trial compares two strategies: standard follow-up with colonoscopy every 18 months versus an approach combining annual liquid biopsies with a colonoscopy every 36 months. The main outcome is the number of new cancer cases diagnosed, confirmed by standard procedures. Secondary outcomes include early cancer detection, lesion identification, diagnostic timing, feasibility, quality of life and healthcare use. Each positive test leads to fast confirmatory exams. The aim is to determine if liquid biopsies can safely reduce invasive procedures while maintaining effective cancer monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Age 35-80
3. Genetically confirmed class 4-5 (likely pathogenic (LP) or pathogenic (P) variant, respectively) in MLH1, MSH2, MSH6, or EPCAM gene.
4. The participant should be insurance covered for the financial costs of the standard surveillance and healthcare related to LS, such as affiliated to Social Security System

Exclusion Criteria:

1. Previously performed proctocolectomy or equivalent (entire colon and rectum removed)
2. Active treatment for cancer within 2 years prior to inclusion.
3. Checkpoint inhibitor therapy within 12 months
4. Pregnancy
5. Participants unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.
6. Persons deprived of their liberty or under protective custody or guardianship.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine whether a multimodal surveillance strategy - using combining concurrent circulating tumor DNA (ctDNA), urine tumor DNA (utDNA), vaginal swab tumor DNA (vsDNA), and stool (qFIT) - is non-inferior to standard-of-care screening surveillance | Baseline, month 12, month 24, month 36, month 48
  Number of newly diagnosed histologically confirmed invasive cancers (CRC, EC, UC) during surveillance and follow-up phases, expressed as cumulative incidence (%) and incidence per 1,000 person-years.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle Colas, Oncogeneticist, Study Director — Institut Curie; Toni Seppala, Surgeon, Study Director — TAMPERE University (Finland)
Locations (9):
- Klinicki Bolnicki Centar Sestre Milosrdnice Ustanova, Zagreb, Croatia
- Masaryk Memorial Cancer Institute, Brno, Czechia
- Tampereen Korkeakoulusäätiö SR, Helsinki, Finland
- GGC Network, Paris, France
- Ist. Tumori di Milano, Milan, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Erasmus Medisch Centrum Rotterdam, Rotterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallon R, Brekelmans C, Martin M, Bours V, Schamschula E, Amberger A, Muleris M, Colas C, Dekervel J, De Hertogh G, Coupier J, Colleye O, Sepulchre E, Burn J, Brems H, Legius E, Wimmer K. Constitutional mismatch repair deficiency mimicking Lynch syndrome is associated with hypomorphic mismatch repair gene variants. NPJ Precis Oncol. 2024 May 24;8(1):119. doi: 10.1038/s41698-024-00603-z. PMID 38789506
- [Background] Wu J, Lin Y, Yang K, Liu X, Wang H, Yu T, Tao R, Guo J, Chen L, Cheng H, Lou F, Cao S, Yu W, Hu H, Ye D. Clinical effectiveness of a multitarget urine DNA test for urothelial carcinoma detection: a double-blinded, multicenter, prospective trial. Mol Cancer. 2024 Mar 19;23(1):57. doi: 10.1186/s12943-024-01974-4. PMID 38504268
- [Background] Willis J, Lefterova MI, Artyomenko A, Kasi PM, Nakamura Y, Mody K, Catenacci DVT, Fakih M, Barbacioru C, Zhao J, Sikora M, Fairclough SR, Lee H, Kim KM, Kim ST, Kim J, Gavino D, Benavides M, Peled N, Nguyen T, Cusnir M, Eskander RN, Azzi G, Yoshino T, Banks KC, Raymond VM, Lanman RB, Chudova DI, Talasaz A, Kopetz S, Lee J, Odegaard JI. Validation of Microsatellite Instability Detection Using a Comprehensive Plasma-Based Genotyping Panel. Clin Cancer Res. 2019 Dec 1;25(23):7035-7045. doi: 10.1158/1078-0432.CCR-19-1324. Epub 2019 Aug 4. PMID 31383735
- [Background] van Liere ELSA, Jacobs IL, Dekker E, Jacobs MAJM, de Boer NKH, Ramsoekh D. Colonoscopy surveillance in Lynch syndrome is burdensome and frequently delayed. Fam Cancer. 2023 Oct;22(4):403-411. doi: 10.1007/s10689-023-00333-4. Epub 2023 May 12. PMID 37171677
- [Background] Moller P, Seppala T, Bernstein I, Holinski-Feder E, Sala P, Evans DG, Lindblom A, Macrae F, Blanco I, Sijmons R, Jeffries J, Vasen H, Burn J, Nakken S, Hovig E, Rodland EA, Tharmaratnam K, de Vos Tot Nederveen Cappel WH, Hill J, Wijnen J, Green K, Lalloo F, Sunde L, Mints M, Bertario L, Pineda M, Navarro M, Morak M, Renkonen-Sinisalo L, Frayling IM, Plazzer JP, Pylvanainen K, Sampson JR, Capella G, Mecklin JP, Moslein G; Mallorca Group (http://mallorca-group.eu). Cancer incidence and survival in Lynch syndrome patients receiving colonoscopic and gynaecological surveillance: first report from the prospective Lynch syndrome database. Gut. 2017 Mar;66(3):464-472. doi: 10.1136/gutjnl-2015-309675. Epub 2015 Dec 9. PMID 26657901
- [Background] Stoffel EM, Murphy CC. Epidemiology and Mechanisms of the Increasing Incidence of Colon and Rectal Cancers in Young Adults. Gastroenterology. 2020 Jan;158(2):341-353. doi: 10.1053/j.gastro.2019.07.055. Epub 2019 Aug 5. PMID 31394082